CLINICAL TRIAL: NCT05503147
Title: A Pharmacological Trial With Sativex® and Gentamicin for Optimized Phamacological Treatment of Older Patients With Focus on Appetite Stimulation and Renal Risk Drugs
Brief Title: Sativex® and Gentamicin for Optimized Pharmagological Treatment in Older Patients (CanPan)
Acronym: CanPan
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ove Andersen (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Regionshospital Nordjylland (Other Government); University of Copenhagen (Other); Region Hovedstadens Apotek (Other Government); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, Research Director and Head of the Department of Clinical Research, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-21044231
Record Dates: First submitted 2022-04-13; First posted 2022-08-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Malnutrition; Anorexia; Cannabis; Aging; Emergency Service, Hospital; Renal Function; Pharmacokinetics
MeSH Terms: conditions — Malnutrition; Anorexia; Marijuana Abuse; Emergencies | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sativex first (blinded) (3 dose of spray) (Experimental): Trial day 1: Sativex (3 dose of spray x 2) Trial day 2: Placebo (3 dose of spray x 2) Trial day 3: Voluntary
  Interventions: Drug: Sativex
- Placebo first (blinded) (3 dose of spray) (Experimental): Trial day 1: Placebo (3 dose of spray x 2) Trial day 2: Sativex (3 dose of spray x 2) Trial day 3: Voluntary
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Sativex® is administered as an oromucosal spray and consists of 2.7 mg tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD) per dosis spray (Cannabis sativa L. extract, cannabis leaf and flower). The dose (3 sprays) is administered twice, at breakfast and lunch, respectively, with approximately 4 hours between each administration.
  Other Names: nabiximols

SUMMARY:
Malnutrition and inappropriate prescribing of renally excreted drugs are common among older persons and are associated with severe consequences such as complicated courses of treatment, mortality, and reduced quality of life. The overall purpose of CanPan is to optimize treatment of older persons with malnutrition with a focus on appetite stimulation and optimized prescribing of renal risk drugs.

The CanPan trial consists of two sub-studies. Substudy 1 will provide knowledge on appetite and appetite stimulation and together, sub study 1 and 2 will offer unique knowledge on how body composition, renal function and biomarkers of organ function influence pharmacokinetics for a highly lipophilic (Sativex®) and hydrophilic (Hexamycin®) drug in older medical patients with malnutrition.

DETAILED DESCRIPTION:
The CanPan trial consists of sub study 1 and sub study 2. Subjects who meet all the inclusion criteria and none of the exclusion criteria are invited to participate in both sub studies. Sub study 1 consist of trial days 1 and 2 and sub study 2 consists of trial day 3.

Sub study 1:

Sub study 1 is a double-blinded, randomized, placebo-controlled, multidose, crossover trial that evaluates the appetite stimulating effect as well as the pharmacokinetics of Sativex®. The primary purpose of sub study 1 is to 1) uncover whether Sativex® has appetite stimulating properties defined as increased energy intake compared to placebo, 2) to develop a pharmacokinetic-pharmacodynamic model, and gain knowledge about the effect of Sativex® on other markers of appetite, the intraocular pressure of the eye and safety parameters.

In sub study 1, subjects receive both Sativex® and placebo. Both Sativex® and placebo are administered as an oromucosal spray. Sativex consists of 2.7 mg tetrahydrocannabinol (THC) and 2.5 mg cannabidiol (CBD) per dose of spray (Cannabis sativa L. extract, cannabis leaf and flower). Subjects receive three dose of spray two times during a trial day. Trial day 1 is planned <14 days after inclusion and there is a 2-week break between trial days 1 and 2 due to a wash-out period. Follow-up visits/phonecalls are made on days 1, 2 and 7 after trial days 1 and 2.

Sub study 2:

Sub-study 2 is a single-dose pharmacokinetic study using gentamicin (Hexamycin®) as a renally excreted model drug. The purpose of sub study 2 is to compare the prediction accuracy of clearance estimates between eGFRpanel (creatinine-cystatinC-beta-2_microglobulin-beta_trace_protein, eGFRcomb (creatinine-cystatinC), eGFRcreatinine (creatinine), uCrCl (24-hour urine creatinine clearance) and mGFR (measured GFR) as covariates in population based pharmacokinetic modeling of gentamicin.

On trial day 3, gentamicin is used as the model substance for a drug that is excreted > 90% renally. Gentamicin is administered as a single dose of 5 mg/kg as an intravenous injection (bolus). The marketed drug, Hexamycin® (40 mg / mL), is used for this purpose. Trial day 3 is held within 4 weeks after trial day 2. Follow-up visits are made on day 1 and 2 after trial day 3.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Admitted to the acute medical department, Hvidovre Hospital
* Can cooperate cognitively and physically (patient reported)
* Low appetite/anorexia of ageing measures by SNAQ score ≤14
* BMI ≤30 (screening)
* Able to read and understand Danish
* Postmenopausal defined as missed periods for at least 12 months before the start of the trial

Exclusion Criteria:

* Regular use of medical cannabis (patient reported)
* Use of medical cannabis within 14 days at baseline (patient reported)
* Recognized or suspected psychotic illness in the subject or the subjects family (medical record and patient report)
* Severe personality disorders (journal)
* Significant psychiatric disorder in addition to mild to moderate depression (medical record)
* Allergy to the ingredients of Sativex®, placebo and Hexamycin® (patient reported)
* Terminal diagnosis (journal)
* Liver transplant (journal)
* Chronic eGFR ≤15 mL / min2 or dialysis treatment (medical record)
* High risk of nephrotoxicity due to existing drug treatment (medical assessment)
* Pacemaker (journal)
* Epilepsy (journal)
* Recurrent seizures (journal)
* Uncontrolled hypertension (journal)
* Food intolerance to the ingredients in the test meals (patient-reported)
* Vegetarian and vegan (patient-reported)
* Unwilling to avoid driving for up to 72 hours after administration of Sativex® (patient-reported)
* Unwilling to avoid alcohol 24 hours up to test days (patient-reported)
* Patients with ascites ( journal)
* Patients with significant edema on the days of the trial (journal / visual inspection)
* In active treatment of cancer or have disseminated cancer (journal)
* Known with brain - or kidney tumor (journal)
* Known with angina pectoris or intermittent claudication
* Known with stroke, AMI, or heart failure (NYHA III-IV) within the past 5 years (journal)
* In isolation
* Obs. Covid-19

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in energy intake (kJ) between Sativex® and placebo | Trial days 1 and 2.
  Measured at test meal
Differences in the objective function value of the population-based pharmacokinetic model when implementing renal clearance assessed by measured GFR (mL/min), or GFR estimates based on different endogenous markers, as covariates on gentamicin clearance | Trial day 3.
  The objective function value (minus two times the log-likelihood) describes the prediction accuracy (goodness-of-fit) of a population pharmacokinetic model. A drop in the objective function value of 6.63 in a model with one (1) added covariate implemented on any specific parameter compared to a base model corresponds to a significant improvement in model fit with a p-value of 0.01 in a chi-squared test.
  Population-based pharmacokinetic modelling is an analysis method performed on pharmacokinetic data, i.e., plasma concentrations over time. Relevant pharmacokinetic parameters are estimated simultaneously by fitting the data to the model. The model structure is found through the analysis and determines which pharmacokinetic parameters are estimated. As a minimum, the clearance and distribution volume of the central compartment are estimated

SECONDARY OUTCOMES:
Differences in the objective function values of the population-based models of CBD and THC when implementing bodyweight, age, and body composition factors as covariates on the pharmacokinetic parameters of the model (e.g., clearance) | Trial days 1 and 2.
  The objective function value (minus two times the log-likelihood) describes the prediction accuracy (goodness-of-fit) of a population pharmacokinetic model. A drop in the objective function value of 6.63 in a model with one (1) added covariate implemented on any specific parameter compared to a base model corresponds to a significant improvement in model fit with a p-value of 0.01 in a chi-squared test.
  Population-based pharmacokinetic-pharmacodynamic modelling is an analysis method performed on pharmacokinetic data, i.e. plasma concentrations over time, coupled to pharmacodynamic data. Relevant pharmacokinetic and -dynamic parameters are estimated simultaneously by fitting the data to the model. The model structure is found through the analysis and determines which pharmacokinetic and -dynamic parameters are estimated. As a minimum, the clearance and distribution volume of the central compartment are estimated
Difference in subjective appetite between Sativex® and placebo | Trial days 1 and 2.
  Using combined subjective appetite scores measured using 100-mm Visual Analogue Scales (VAS), with 0.0 as the minimum value and 10.0 as the maximum value. The following will be used to calculate a combined appetite score: [desire to eat + hunger + prospective food consumption + (10.0 - fullness) + (10.0 - satiety)], with higher scores indicating better appetite.
Differences in the appetite hormones, total ghrelin and glucagon like peptide 1 (GLP-1) between Sativex® and placebo | Trial days 1 and 2.
  The appetite hormones (total ghrelin, GLP-1) is measured from blood samples
Change in the intraocular pressure of the eye between Sativex® and placebo | Trial days 1 and 2.
  Measured by Icare ic100 tanometer
Safety parameter (CNS effects) for Sativex® | Trial days 1 and 2.
  Measured using 100-mm Visual Analogue Scales (VAS), with 0.0 as the minimum value and 10.0 as the maximum value. Higher scores indicate a larger effect.
Safety parameter (cognition) for Sativex® | Trial days 1 and 2.
  Measured using Hopkins Verbal Learning Test-Revised for a total score of the following sub-tests: 'Total recall', 'Delayed recall', 'Retention' and 'Recognition'. Higher scores indicate better performance.
Safety parameter (balance disorders) for Sativex® | Trial days 1 and 2.
  Bergs Balance Test is used to measure balance disorders. Balance disorders are defined as a summerated score of ≤45.
Safety parameter (blood pressure) for Sativex® | Trial days 1 and 2.
  Blood pressure is measured in millimeter of mercury (mmHg) using automatic standardized equipment.
Safety parameter (heart rate) for Sativex® | Trial days 1 and 2.
  Heart rate is measured in beats per minute (bpm) using automatic standardized equipment.
Correlation coefficient between clearance of gentamicin and clearance determined as mGFR or eGFR | Trial day 3.
  Pharmacokinetic modeling
Change in plasma creatinine µmol/L between baseline and 22 hours after administration of gentamicin | Trial day 3
  Changes in kidney biomarkeres before and after administration of gentamicin
Change in plasma cystatin C mg/L between baseline and 22 hours after administration of gentamicin | Trial day 3
  Changes in kidney biomarkers before and after administration of gentamicin
Change in plasma NGAL ng/mL between baseline and 22 hours after administration of gentamicin | Trial day 3
  Changes in kidney biomarkers before and after administration of gentamicin
Change in plasma KIM-1 pg/mL between baseline and 22 hours after administration of gentamicin | Trial day 3
  Changes in kidney biomarkers before and after administration of gentamicin

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, Study Chair — Hvidovre University Hospital; Rikke L Nielsen, Study Chair — Hvidovre University Hospital
Locations (1):
- Clinical Research Centre, Hvidovre, Denmark

REFERENCES:
- [Derived] Nielsen RL, Bornaes O, Christensen LWS, Juul-Larsen HG, Storgaard IK, Kallemose T, Jorgensen LM, Jawad BN, Altintas I, Lund TM, Rasmussen HH, Munk T, Andersen O, Houlind MB, Andersen AL. The appetite stimulating effect and safety of delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) in older patients with poor appetite: A triple-blinded, randomized, placebo-controlled, cross-over trial. Clin Nutr. 2025 Apr;47:248-257. doi: 10.1016/j.clnu.2025.02.024. Epub 2025 Feb 24. PMID 40069983